CLINICAL TRIAL: NCT03885869
Title: Investigation of Relationships Between Joint Position Sense, Plantar Sensation, Balance and Dual Task Performance in Individuals With Type 2 Diabetes
Brief Title: Joint Position Sense, Plantar Sensation, Balance and Dual Task Performance in Individuals With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Assistant Professor, Ankara Yildirim Beyazıt University
Other Study IDs: 2019-83
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes Mellitus; Balance
Keywords: Type 2 Diabetes Mellitus; Joint Position Sense; Plantar Sensation; Balance; Dual Task Performance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetics: Type 2 diabetic individuals aged 30-65 years
  Interventions: Other: Ankle Joint Position Sensation Evaluation; Other: Knee Joint Position Sensation Evaluation; Other: The Evaluation of Plantar Sensation; Other: The Evaluation of Balance; Other: Evaluation of Dual Task Performance; Other: General Evaluation Form

INTERVENTIONS:
Other: Ankle Joint Position Sensation Evaluation — In this test, individuals are placed in the supine position with their eyes closed for prevent visual cues; measurements are performed with the plex of the goniometer, 1.5 cm below the lateral malleol, the fixed arm parallel to the long axis of the fibula and the movable arm parallel to the long axis of the 5th metatarsal. Desired target angles were defined as 10 ° dorsi flexion, 10 ° plantar flexion and 20 ° plantar flexion. Individuals are instructed to focus on the position of the ankle joints in space for 5 s by bringing the feet in neutral position to the target position by the researcher. This procedure is repeated 3 times and the patient is expected to learn this position. The target angle is then asked to repeat in the testing phase. The measurement is repeated 3 times for each target angle. As a result criterion; By recording the absolute value of the deviation amounts from the target angles; The averages of the deviations during the 3 repetitions are averaged.
Other: Knee Joint Position Sensation Evaluation — Bilateral knee joint position sensation will be evaluated in the literature with an analogue inclinometer(BASELINE®),which is a valid and reliable method for measuring joint position sensations.Measurements were planned to made in the sitting position,with the eyes of the individual closed and the joint to be evaluated bare,without any socks or shoes worn,fixing the inclinometer with a strap to the lower leg perpendicular to the knee flexion axis.In this measurement,the knees of the participants are passively shifted from the initial (90°flexion)position to the 30°flexion position,at this point 5 sec is waited and after they are told to keep this angle in mind,the starting position is returned.This procedure is repeated 3 times and the patient is expected to learn this position.After the individuals are rested for 5 s,they are asked to actively perform the target angle again.The same procedure was planned to be repeated 3 times for each angle at 45° and 60° knee flexion target angles.
Other: The Evaluation of Plantar Sensation — In the plantar sensory evaluation of the participants, Semmes-Wenstein Monofilament, which is frequently used in the literature and to be a reliable method in the diagnosis of neuropathy, was aimed to be tested by touching 7 regions on the foot base .
  In this evaluation, the individual is in the supine position, the physiotherapist is at the foot end of the patient; monofilament should be applied 90⁰ to the surface.
  The filament thickness which is the first feeling of the individual is recorded by being asked whether the individual is feeling. The 3 most commonly used monofilaments for patients with diabetic neuropathy are 4.17, 5.07 and 6.10 monofilaments. The highest monofilament value is the hardest and most difficult bending monofilament.
Other: The Evaluation of Balance — In order to evaluate the static and dynamic balances of the participants, determination of open and closed postural oscillations and stability limits were planned with Prokin branded isokinetic balance system.
Other: Evaluation of Dual Task Performance — In order to evaluate double task performances, it is planned to evaluate 1 dynamic and 1 static 2 different performances, including Time Up and Go Test (TUG) and single leg standing time. For each performance; the single task, the motor second task and cognitive seconder tasks separately, and again for each application to be performed in such a way that two trials, the average time was planned to record. Motor and cognitive tasks for each test are planned as described below.
  Motor Task (TUG): Carrying cup full of water on tray. Cognitive Task (TUG): Counting the days of the week backwards from the current day Motor Task (Single Leg Standing Time): Hand-Over ball transfer Cognitive Task (Single Leg Standing Time): Counting backward month names from the current month
Other: General Evaluation Form — A form, which is prepared by us, including demographic information and physical characteristics of the individuals.

SUMMARY:
Diabetes is a chronic disease characterized by hyperglycemia, which occurs when insulin is inadequate or the body's produced insulin cannot be used effectively, but according to the World Health Organization 2016 Global Report on Diabetes, it is an important public health problem that is one of the four priority non-infectious diseases. In addition to high mortality rates caused by diabetes-related complications, it is known that it can cause low quality of life and many additional problems in individuals. These complications and damage, which may be caused by diabetes, may result in reduced blood flow combined with neuropathy; As a result, foot ulcers, infections and consequently the need for amputation may increase. In addition to the additional complications caused by diabetic neuropathy, protective plantar sensory loss and decreased joint position have been reported in the literature. In particular, investigators did not find any comprehensive studies examining the relationship between these sensory changes and the dual task performance in diabetic subjects. In this study, investigators aimed to investigate the relationship between joint position sense, plantar sensation, balance and dual task performance in individuals with type 2 diabetes and to contribute to the literature with evidence-based, objective results.

DETAILED DESCRIPTION:
The aim of this study is to investigate that the relationships between joint position sensation, plantar sensation, balance and dual task performance in type 2 diabetic patients.

First of all, a general evaluation form including demographic information and physical characteristics of the individuals who voluntarily agree to participate in the study and approve the informed consent form, will be filled. Then, with the first findings to be obtained, determination of sample size was planned. Bilateral ankle joint position sensation with goniometer, bilateral knee joint position sensation with an analog inclinometer (BASELINE® Bubble inclinometer-USA), plantar sensation with Semmens-Wenstein monofilaments, equilibrium with Prokin Isokinetic Balance System, dual task performance will be evaluated with adding motor and cognitive secondary tasks to the Time Up and Go Test and single leg balance tests.

ELIGIBILITY:
Inclusion Criteria:

* to accept to participate in the study voluntarily,
* to being diagnosed with type 2 diabetes,
* to being 30-65 age range.

Exclusion Criteria:

* refuse to participate in the study,
* Not cooperating,
* Being orthopedic, neurological and any other systemic disease,
* Being pregnant,
* Loss of vision,
* Loss of hearing,
* To be a standing diabetic ulcer,
* A Mini Mental Test score of 23 or less.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic individuals between the ages of 30-65
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
The Evaluation of Ankle Joint Position Sensation | 1 month
  In this test, individuals are placed in the supine position with their eyes closed for prevent visual cues; measurements are performed with the plex of the goniometer, 1.5 cm below the lateral malleol, the fixed arm parallel to the long axis of the fibula and the movable arm parallel to the long axis of the 5th metatarsal. Desired target angles were defined as 10 ° dorsi flexion, 10 ° plantar flexion and 20 ° plantar flexion. Individuals are instructed to focus on the position of the ankle joints in space for 5 s by bringing the feet in neutral position to the target position by the researcher. This procedure is repeated 3 times and the patient is expected to learn this position. The target angle is then asked to repeat in the testing phase. The measurement is repeated 3 times for each target angle. As a result criterion; By recording the absolute value of the deviation amounts from the target angles; The averages of the deviations during the 3 repetitions are averaged.
The Evaluation of Knee Joint Position Sensation | 1month
  Bilateral knee joint position sensation will be evaluated in the literature with an analogue inclinometer(BASELINE®),which is a valid and reliable method for measuring joint position sensations.Measurements were planned to made in the sitting position,with the eyes of the individual closed and the joint to be evaluated bare,without any socks or shoes worn,fixing the inclinometer with a strap to the lower leg perpendicular to the knee flexion axis.In this measurement,the knees of the participants are passively shifted from the initial(90°flexion)position to the 30°flexion position,at this point 5 sec is waited and after they are told to keep this angle in mind,the starting position is returned.This procedure is repeated 3 times and the patient is expected to learn this position.After the individuals are rested for 5 s,they are asked to actively perform the target angle again.The same procedure was planned to be repeated 3times for each angle at 45° and 60°knee flexion target angles.
The Evaluation of Plantar Sensation | 1month
  In the plantar sensory evaluation of the participants, Semmes-Wenstein Monofilament, which is frequently used in the literature and to be a reliable method in the diagnosis of neuropathy, was aimed to be tested by touching 7 regions on the foot base .
  In this evaluation, the individual is in the supine position, the physiotherapist is at the foot end of the patient; monofilament should be applied 90⁰ to the surface.
  The filament thickness which is the first feeling of the individual is recorded by being asked whether the individual is feeling. The 3 most commonly used monofilaments for patients with diabetic neuropathy are 4.17, 5.07 and 6.10 monofilaments. The highest monofilament value is the hardest and most difficult bending monofilament.
Evaluation of Balance Performance | 1month
  In order to evaluate the static and dynamic balances of the participants, determination of open and closed postural oscillations and stability limits were planned with Prokin branded isokinetic balance system.
The Evaluation of Dual Task Performance | 1month
  In order to evaluate double task performances, it is planned to evaluate 1 dynamic and 1 static 2 different performances, including Time Up and Go Test (TUG) and single leg standing time. For each performance; the single task, the motor second task and cognitive seconder tasks separately, and again for each application to be performed in such a way that two trials, the average time was planned to record. Motor and cognitive tasks for each test are planned as described below.
  Motor Task (TUG): Carrying cup full of water on tray. Cognitive Task (TUG): Counting the days of the week backwards from the current day Motor Task (Single Leg Standing Time): Hand-Over ball transfer Cognitive Task (Single Leg Standing Time): Counting backward month names from the current month.

CONTACTS AND LOCATIONS:
Overall Officials: Nazire Nur Yıldız, PT, Principal Investigator — AYBU Institute of Health Sciences Department of Physiotherapy and Rehabilitation Master Program/Master Degree Student
Locations (1):
- Ankara Yıldırım Beyazıt University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No